CLINICAL TRIAL: NCT03654261
Title: 1-Day Cognitive Behavioural Therapy Workshops for Postpartum Depression
Brief Title: 1-Day CBT Workshops for PPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Ryan Van Lieshout, MD, PhD, Assistant Professor, Department of Psychiatry and Behavioural Neurosciences, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1Day-CBT
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Postpartum Depression
Keywords: Cognitive Therapy; Workshop; Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1-Day CBT Workshop - Immediate (Experimental): Women assigned to the immediate workshop group will participate in the first of two workshops (9 weeks apart).
  Interventions: Behavioral: Cognitive Behavioural Therapy
- 1-Day CBT Workshop - Waitlist (Experimental): Women assigned to the waitlist will participate in the second of two workshops (12 weeks apart).
  Interventions: Behavioral: Cognitive Behavioural Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy — The intervention is a 1-day Cognitive Behavioural Therapy based workshop.

SUMMARY:
Postpartum depression (PPD) affects up to 20% of women and has profound effects on women and their families. Clinical practice guidelines recommend that the majority of women with PPD receive psychotherapy. A previously validated 1-day CBT workshop has been adapted for depression for use with women experiencing PPD and living in the community. 476 women will be randomized to active treatment or a 12 week wait list in each setting and compare changes in depression, mother-infant attachment, service utilization, quality of life, and offspring behaviour.

DETAILED DESCRIPTION:
Postpartum depression (PPD) affects up to 20% of women and has profound effects on women and their families (1,2). Indeed, the cost of one case of PPD is estimated to exceed $150,000 (3). Unfortunately, fewer than 15% of women with PPD receive evidence-based care (4), which is at least partly due to difficulties accessing treatment, particularly therapies that are most preferred (e.g., psychotherapy (5)).

Clinical practice guidelines recommend that the majority of women with PPD receive psychotherapy (e.g., cognitive behavioural therapy (CBT)) as a 1st-line treatment (6). Moreover, consensus recommendations such as those made by the US Preventive Services Task Force suggest that screening only occur in settings where evidence-based counselling such as CBT is readily available (7). In order to increase access to treatment, screening efforts have been undertaken by public health units province-wide in Ontario. This has occurred despite the widespread availability of evidence-based psychotherapies.

A previously validated 1-day CBT workshop has been adapted for depression for use with women experiencing PPD and living in the community. 476 women will be randomized to active treatment or a 12 week wait list in each of 5 settings (Simcoe County, Kitchener-Waterloo Region, Halton Region, Prince Edward County, Elgin County), and compare changes in depression, mother-infant attachment, service utilization, quality of life, and offspring behaviour.

If this intervention is eventually proven effective, more women would receive treatment and the burden of PPD on women, families, and the healthcare system would be significantly reduced. Providing women with PPD with CBT skills at this crucial stage in life also has the capacity to prevent future depressive relapse with significant benefits for patients, families, employers, and the healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* infant <12 months
* 18 years or older
* EPDS score >10

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 461 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-08-17 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale (EPDS) | 3 months
  EPDS is the 10-item gold standard measure of PPD. A score >10 is consistent with PPD and changes in scores >4 are accepted as being indicative of clinically significant change
Beck Depression Inventory-II | 3 months
  The Beck Depression Inventory is a 21-item scale that assesses the emotional and cognitive symptoms of depression as the EPDS does, but additionally captures the somatic symptoms of depression. Higher scores on the BDI-II indicate more sever depression. The minimum score is 0 and maximum score is 63. Items are summed to generate a total score. 0-13 = minimal depression; 14-19 = mild depression; 20-28 = moderate depression; 29-63 = severe depression.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder-7 (GAD-7) | 3 months
  The GAD-7 is a 7-item self-report scale that taps generalized anxiety disorder, the most common comorbidity of PPD. The minimum score is 0 and the maximum score is 21. Items are summed to generate a total score. Scores of 5-9 indicate mild anxiety, 10-14 indicate moderate anxiety and 15 or greater indicate severe anxiety.
Postpartum Bonding Questionnaire | 3 months
  Postpartum Bonding Questionnaire is a 25-item maternal report scale that is designed to detect disorders of the mother-infant relationship. Scores range on each question from 0 (Always) to 5 (Never) and are summed to generate subscale scores. The subscales include: impaired bonding, rejection and pathological anger, infant focused anxiety and incipient abuse. Higher scores indicate problems with bonding.
Client Satisfaction Questionnaire | Immediately after workshop
  The Client Satisfaction Questionnaire (CSQ-8) is an 8-item patient reported scale that is designed to measure client satisfaction with services. The Maximum score is 32 and the minimum score is 4. Higher scores indicate greater satisfaction.
Healthcare Utilization | 3 months
  As depression is associated with increased rates of healthcare use, mothers will answer the Health Care Utilization questions of the Canadian Community Health Survey at all time points. Mothers will also answer the General Help-Seeking Questionnaire and the Mental Help Seeking Intention Scale at all time points, in order to measure the likelihood that they will seek help from healthcare professionals.
Infant Behaviour Questionnaire-Revised (Very short form) | 3 months
  To assess infant temperament if infants. The measure takes a mean value of the questions to which a response was provided.
Strengths and Difficulties Questionnaire | 3 months
  To assess temperament of 2-4 year olds. Each response has values of 0, 1 and 2. These are summed to generate a total score for each subscale: Emotional Problems Scale, Conduct Problems Scale, Hyperactivity Scale, Peer Problems Scale, Prosocial Scale. The minimum score for each scale is 0 and the maximum is 10. Higher scores indicate greater difficulties.
Early Childhood Behaviour Questionnaire (very short form) | 3 months
  To assess temperament of children 18-36 months. The subscales include negative affect, surgency and effortful control. The measure takes a mean value of the questions to which a response was provided.
EQ-5D | 3 months
  The EQ-5D, a measure of health-related quality of life will also be completed by mothers. Health status is measured on five dimensions on three-point scales. The associated tariffs for Canada are then applied to calculate quality-adjusted life-years (QALYs). The instrument also includes a visual analogue scale, allowing individuals to rate their current health status on a scale from 0 (worst) to 100 (best).

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Van Lieshout, MD, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Layton H, Owais S, Savoy CD, Van Lieshout RJ. Depression, Anxiety, and Mother-Infant Bonding in Women Seeking Treatment for Postpartum Depression Before and During the COVID-19 Pandemic. J Clin Psychiatry. 2021 Jul 6;82(4):21m13874. doi: 10.4088/JCP.21m13874. PMID 34232578